CLINICAL TRIAL: NCT05424107
Title: Nutritional Status of South Spanish Children: A Mediterranean Diet Nutritional Intervention of Children With Insulin Resistance From a Rural Area
Brief Title: A Mediterranean Intervention on Prediabetic Children
Acronym: INTKIDMEDPRED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pilar Aparicio Martinez (Other)
Collaborators: Instituto Maimónides de Investigación Biomédica de Córdoba (IMIBIC) (Unknown)
Responsible Party: Sponsor-Investigator, Pilar Aparicio Martinez, Researcher and Lecture at the University and IMIBIC, Universidad de Córdoba
Organization: Universidad de Córdoba (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2353; 251 (Other: PEIBA)
Record Dates: First submitted 2022-06-09; First posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Prediabetic State
Keywords: Nutritional intervention; Prediabetes; Children; Mediterranean diet
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: This is a study with pre-and post-intervention evaluation, randomized intervention in parallel groups EG and CG, in schoolchildren with analytical data of pre-diabetes. The study design was divided into two phases. In each phase, a follow-up was carried out with five visits, from the initial visit (v0) to the final visit (v4).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-nutritional intervention (Experimental): Children with a prediabetic status that followed up the sessions without nutritional intervention by a health care professional
  Interventions: Other: KIDMED

INTERVENTIONS:
Other: KIDMED — Pre-and post-intervention evaluation of the adherence to the Mediterranean diet and its effect on prediabetic state, as well as, other anthropometric values.

SUMMARY:
Prediabetes is a pathological condition where the blood glucose concentration is higher than normal concentrations but lower than those considered in type 2 diabetes mellitus (DM2) diagnosis. Until a few years ago, this prediabetes occurred in adults with associated risk factors such as being overweight or obese, sedentary lifestyle, poor eating habits, and cardiovascular problems, among others. Recently, it has begun to be detected in children, with family eating habits becoming more critical. Therefore, the objectives of this study were to determine the efficacy of the nutritional intervention in children with analytical data on pre-diabetes; and the secondary ones proposed were to evaluate if an individualized and directed nutritional intervention compared to the standardized one supposes an improvement in children's dietary habits and to determine if nutritional education improves anthropometric parameters and adherence to a Mediterranean diet, through the evaluation of the Mediterranean Diet Quality Index (KIDMED).

ELIGIBILITY:
Inclusion Criteria:

* Presence of HbA1c levels between 5.7 and 6.4% in the blood tests
* Signed informed consent by the minor
* Signed informed consent by the minor's parents or guardians.

Exclusion Criteria:

* Presence of HbA1c levels below 5.7%
* Presence of HbA1c levels above 6.4%
* Presence of pathological metabolic diseases, such as diabetes or metabolic syndrome
* Lack of the signed informed consent by the minor and legal guardian

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 254 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2020-01-04 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
HbA1c levels | Up to six months
  The HbA1c were measured at the initial visit (V0) and during the last visit (V4)

SECONDARY OUTCOMES:
Height (m2) | Up to six months
  The height of the children was measured via the Omron BF-511 impedance mete, being classified to Melo Sailor's tables of child growth. The measure of the impedance was taken at the initial visit (V0) and at the last visit (V4)
Weight (kg) | Up to six months
  The weight (kg) of the children was measured via the Omron BF-511 impedance mete, being classified to Melo Sailor's tables of child growth. The measure of the impedance was taken at the initial visit (V0) and at the last visit (V4)
Waist circumference (cm) | Up to six months
  The waist circumference (cm) of the children was measured via an inextensible measuring tape at the initial visit (V0) and at the last visit (V4)
Hip circumference(cm) | Up to six months
  The hip circumference(cm) of the children was measured via an inextensible measuring tape at the initial visit (V0) and at the last visit (V4)
Arm circumference (cm) | Up to six months
  The arm circumference (cm) of the children was measured via an inextensible measuring tape at the initial visit (V0) and at the last visit (V4). The measurement follows the recommendations of the International Standards for Anthropometric Assessment
Body mass index (kg/m2) | Up to six months
  The children's body mass index (kg/m2) was obtained following the World Health Organization's recommendations and guidelines, being classified to Melo Sailor's tables of child growth. The calculation of the BMI was obtained at the initial visit (V0) and the last visit (V4)
Validated nutritional assessment questionnaire: adherence to the Mediterranean diet (KIDMED) | Up to six months
  The KIDMED was used to determine adherence to the change in diet from the initial visit (V0) and the final visit (V4). This questionnaire is formed by 16 questions related to adherence to the Mediterranean diet, in addition to 7 items complementary to the test. All questions were answered positively or negatively. Of the 16 main questions, questions number 6, 11, 14, and 16, in their affirmative answers had a negative meaning, so they were worth (-1), on the other hand, the remaining questions whose affirmative answers represented a positive value concerning the Mediterranean diet were scored with (+1). Negative responses do not score (0). According to the test, the results are grouped into different levels of adherence to the Mediterranean diet, low (score 0 to 3), medium (score 4-7), and high (8 to 12).
The Food Frequency Questionnaire (FFQ) | Up to six months
  The Food Frequency Questionnaire (FFQ) was used to determine the consumption of food and the change in diet from the initial visit (V0) and the final visit (V4). The Food Frequency Questionnaire (FFQ) includes 137 foods classified into 14 food groups (dairy products, eggs, meat or meat products, fish or shellfish, vegetables, potatoes, fruits, nuts, legumes, cereals, olive oil, pastries, cakes or sweets, and alcoholic beverages). Frequencies are recorded using a 9-category Likert-type scale (from "rarely" to "6 or more times per day"). In addition, the consumption of common foods in this population group was collected, such as juices (nectars, concentrates, etc.), sweets or sugary breakfast cereals (with chocolate, honey, etc.), and the techniques habitual culinary used in the houses. Energy and nutrient intakes were calculated using Spanish food composition tables
Decalogue of healthy eating | Up to six months
  The decalogue of healthy eating was used to analyze the healthy eating habits and the change in diet from the initial visit (V0) and the final visit (V4). This survey was developed for the internal control of adherence to the prescribed dietary recommendations, is a tool that has allowed the dietitian and the children/parents to know which were the dietary aspects to improve quickly and simple; according to the test it was grouped into different levels of adherence to the diet, low (score 0 to 3), medium (score 4-7) and high (8 to 10).

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Fonseca del Pozo, PhD, Principal Investigator — Maimónides Biomedical Research Institute of Córdoba
Locations (1):
- Ayuntamiento de Pedra Abad, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Undecided
We have decided to first present the data in different forums and journals before making the database available